CLINICAL TRIAL: NCT03624647
Title: An 8-Week Clinical Comparison of an Experimental Power Brush Compared to a Manual Toothbrush in the Reduction of Gingivitis and Plaque
Brief Title: A Clinical Comparison of an Experimental Power Brush Compared to a Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018030
Record Dates: First submitted 2018-08-06; First posted 2018-08-10 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Gingivitis; Dental Plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Power toothbrush (Experimental)
  Interventions: Device: Power toothbrush
- Manual toothbrush (Placebo Comparator)
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Power toothbrush — Experimental power toothbrush
  Arms: Power toothbrush
Device: Manual toothbrush — Marketed manual toothbrush
  Arms: Manual toothbrush

SUMMARY:
The objective of the study is to evaluate and compare the efficacy of an experimental power brush to a regular manual brush in the reduction of gingivitis and dental plaque over an 8 week period by using the Modified Gingival Index, the Gingival Bleeding Index and the Rustogi Modification of the Navy Plaque Index.

ELIGIBILITY:
Inclusion Criteria:

* give written informed consent prior to study participation and be given a signed copy of their informed consent form
* be at least 18 years of age and typically use a manual toothbrush;
* be in good general health as determined by the investigator/designee based on a review/update of their medical history;
* possess a minimum of 16 natural teeth with facial and lingual scorable surfaces;
* have a Baseline pre-brushing MGI score of at least 1.75;
* have a Baseline pre-brushing RMNPI score of greater than 0.5;
* have at least 20 bleeding sites (sites with a score of 1 or 2 on the GBI index) for Baseline pre-brushing;
* agree not to participate in any other oral care study for the duration of this study;
* agree to not to have any elective dentistry, including dental prophylaxis, until study completion and to report any non-study dentistry received at any time during the course of this study;
* agree to refrain from using any non-study oral hygiene products for the study duration;
* agree to return for all their scheduled visits and to follow all study procedures;
* refrained from brushing their teeth or from performing any other oral hygiene procedures anytime within the 12 hours prior to their morning brushing and agree to follow these same restrictions prior to all visits except (the Week 1 p.m. visit);
* refrained from any oral hygiene, eating, drinking* (except small sips of water), chewing gum, and tobacco use for at least 3 hours but not more than 6 hours prior to this visit and agree to follow these same restrictions prior to all p.m. visits.

Exclusion Criteria:

* a condition requiring the need for antibiotic premedication prior to dental procedures;
* severe periodontal disease, including but not limited to, purulent exudates, generalized mobility, and/or severe recession;
* teeth that are grossly carious, fully crowned, or extensively restored;
* active treatment for the following conditions: periodontitis, cancer, or a seizure disorder;
* report to be nursing or pregnant, or intend to become pregnant any time during the course of this study;
* taking an antibiotic or using a chlorhexidine mouth rinse any time within the previous 2 weeks;
* have any of the following: orthodontic appliances, removable partial dentures, peri/oral piercings, a pacemaker or other implanted device;
* oral/gum surgery within the previous two months;
* a disease or condition that could possibly interfere with examination/procedures or with the subject's safe completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index | Baseline
  MGI is a validated assessment of Gingival inflammation using a 4 point range where 0 (absence of inflammation) to 4 (severe inflammation).
Modified Gingival Index | Week 1
  MGI is a validated assessment of Gingival inflammation using a 4 point range where 0 (absence of inflammation) to 4 (severe inflammation).
Modified Gingival Index | Week 8
  MGI is a validated assessment of Gingival inflammation using a 4 point range where 0 (absence of inflammation) to 4 (severe inflammation).
Rustogi Modification of the Navy Plaque Index | Baseline
  RMNPI is a validated assessment of visual surface dental plaque using a dichotomous scale 0 (absence) to 1 (presence).
Rustogi Modification of the Navy Plaque Index | Week 1
  RMNPI is a validated assessment of visual surface dental plaque using a dichotomous scale 0 (absence) to 1 (presence).
Rustogi Modification of the Navy Plaque Index | Week 8
  RMNPI is a validated assessment of visual surface dental plaque using a dichotomous scale 0 (absence) to 1 (presence).

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research Ltd., Mississauga, Ontario, Canada